CLINICAL TRIAL: NCT01894191
Title: A Randomized, Controlled Trial Comparing the Adenoma Detection Rate With Air Insufflation, Water Immersion and Water Exchange During Colonoscopy
Brief Title: Comparing the Adenoma Detection Rate With Air Insufflation, Water Immersion and Water Exchange
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalin Tzu Chi General Hospital (Other)
Collaborators: Sepulveda Ambulatory Care Center, VAGLAHS (Unknown)
Responsible Party: Principal Investigator, Yu-Hsi hsieh, Doctor, Dalin Tzu Chi General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DalinTCGH-hsieh-03
Record Dates: First submitted 2013-07-03; First posted 2013-07-10 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Adenoma
Keywords: adenoma detection rate; colonoscopy; water exchange
MeSH Terms: conditions — Adenoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- air insufflation (Active Comparator): Air insufflation will be used throughout whole procedure of colonoscopy
  Interventions: Procedure: Air insufflation
- water immersion (Active Comparator): Water will be infused during the insertion phase and removed during withdrawal phase of colonoscopy.
  Interventions: Procedure: water immersion
- water exchange (Active Comparator): Water will be infused and removed during insertion phase of colonoscopy
  Interventions: Procedure: Water exchange

INTERVENTIONS:
Procedure: Air insufflation — Insufflation during colonoscopy including insertion phase
  Arms: air insufflation
Procedure: water immersion — Water will infused during insertion phase and removed during withdrawal phase of colonoscopy
  Arms: water immersion
Procedure: Water exchange — Water will infused and removed during insertion phase of colonoscopy
  Arms: water exchange

SUMMARY:
Interval (missed) cancers and lower than expected mortality reduction of proximal colon cancers in the United States and elsewhere after screening colonoscopy drew attention to quality indicators. Missed adenomas which are more likely to be in the proximal colon may be contributing factors. An independent predictor of the risk of interval cancers is adenoma detection rate. In pilot observations, the investigators showed that water exchange enhanced adenoma detection in the right colon (cecum to hepatic flexure). This prospective, randomized controlled trial will compare water exchange with water immersion and traditional air insufflation in patients undergoing colonoscopy. The investigators test the hypothesis that compared with air insufflation and water immersion, water exchange produces a significantly higher adenoma detection rate in the right colon.

DETAILED DESCRIPTION:
All of the procedures will be recorded and stored as digital files.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing colonoscopy performed by the participating endoscopists

Exclusion Criteria:

* obstructive lesions of the colon known before colonoscopy
* massive ascites
* past history of partial colectomy
* refusal to provide written informed consent

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 651 (Actual)
Dates: Start 2013-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
adenoma detection rate | one week

SECONDARY OUTCOMES:
adenoma detection rate in proximal colon | one week
  the proportion of patients with the presence of adenoma in the proximal colon

OTHER OUTCOMES:
post-procedure discomfort and 30 days complication rate | 30 days
  telephone follow up for post-procedure discomfort and 30 days complication rate

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Hsi Hsieh, MD, Principal Investigator — Buddhist Dalin Tzu Chi Hospital
Locations (2):
- Sepulveda Ambulatory Care Center, Veterans Affairs Greater Los Angeles Healthcare System, North Hills, California, United States
- Dalin Tzu Chi General Hospital, Chiayi City, Taiwan, Taiwan

REFERENCES:
- [Background] Bressler B, Paszat LF, Vinden C, Li C, He J, Rabeneck L. Colonoscopic miss rates for right-sided colon cancer: a population-based analysis. Gastroenterology. 2004 Aug;127(2):452-6. doi: 10.1053/j.gastro.2004.05.032. PMID 15300577
- [Background] Stock C, Pulte D, Haug U, Brenner H. Subsite-specific colorectal cancer risk in the colorectal endoscopy era. Gastrointest Endosc. 2012 Mar;75(3):621-30. doi: 10.1016/j.gie.2011.10.025. PMID 22341107
- [Background] Leung FW, Amato A, Ell C, Friedland S, Harker JO, Hsieh YH, Leung JW, Mann SK, Paggi S, Pohl J, Radaelli F, Ramirez FC, Siao-Salera R, Terruzzi V. Water-aided colonoscopy: a systematic review. Gastrointest Endosc. 2012 Sep;76(3):657-66. doi: 10.1016/j.gie.2012.04.467. PMID 22898423
- [Background] Radaelli F, Paggi S, Amato A, Terruzzi V. Warm water infusion versus air insufflation for unsedated colonoscopy: a randomized, controlled trial. Gastrointest Endosc. 2010 Oct;72(4):701-9. doi: 10.1016/j.gie.2010.06.025. PMID 20883846
- [Background] Hsieh YH, Lin HJ, Tseng KC. Limited water infusion decreases pain during minimally sedated colonoscopy. World J Gastroenterol. 2011 May 7;17(17):2236-40. doi: 10.3748/wjg.v17.i17.2236. PMID 21633535
- [Derived] Hsieh YH, Tseng CW, Hu CT, Koo M, Leung FW. Prospective multicenter randomized controlled trial comparing adenoma detection rate in colonoscopy using water exchange, water immersion, and air insufflation. Gastrointest Endosc. 2017 Jul;86(1):192-201. doi: 10.1016/j.gie.2016.12.005. Epub 2016 Dec 15. PMID 27988288